CLINICAL TRIAL: NCT01616576
Title: Evaluation of a HiRes™ Optima Sound Processing Strategy for the HiResolution™ Bionic Ear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Bionics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR0611
Record Dates: First submitted 2012-06-01; First posted 2012-06-12 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2014-08

CONDITIONS: Severe to Profound Hearing Loss; in Adult Users of Advanced Bionics HiResolution™ Bionic Ear System
Keywords: cochlear implant; adults; HiResolution™; Fidelity 120™; listening benefits; noise; cochlear implant benefit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control first, then Experimental (Group A) (Experimental): Initial subject use of Control Sound Processing Strategy for the first week, followed by subject use of Experimental (HiRes™ Optima) Sound Processing Strategy for the HiResolution™ Bionic Ear System for the second week.
  Interventions: Device: Control first, then Experimental
- Experimental first, then Control (Group B) (Experimental): Initial subject use of Experimental (HiRes™ Optima) Sound Processing Strategy for the first week for the HiResolution™ Bionic Ear System, followed by subject use of the Control Sound Processing Strategy for the second week.
  Interventions: Device: Experimental first, then Control

INTERVENTIONS:
Device: Control first, then Experimental — Control condition is currently marketed sound processing strategy.
  Arms: Control first, then Experimental (Group A)
Device: Experimental first, then Control — Experimental condition is newly modified sound processing strategy.
  Arms: Experimental first, then Control (Group B)

SUMMARY:
The purpose of this study is to compare a new sound processing strategy to the current sound processing strategy.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral user of CII/HiRes90K™ implant(s) (minimum of one year in each implanted ear), Harmony™ BTE processor(s) with HiRes Fidelity 120™ (with or without ClearVoice™) as preferred sound processing strategy
* 18 years of age or older at time of implant
* Postlingual onset of severe-to-profound hearing loss (≥ 6 years of age)
* At least moderate open-set speech recognition abilities (defined as CNC word score ≥ 50% in medical records or assessed at the Baseline Visit with implant alone for unilateral users, with both implants together for bilateral users)
* English language proficiency
* Willingness to use a Harmony™ BTE processor and refrain from ClearVoice™ use for the duration of the study
* Willingness and ability to participate in all scheduled procedures outlined in the protocol

Exclusion Criteria:

• Presence of any additional disabilities that would prevent or interfere with participation in the required speech perception testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - House Ear Clinic, Los Angeles, California
  - Tampa Bay Hearing and Balance, Tampa, Florida
  - Carle Clinic Association, Urbana, Illinois
  - Midwest Ear Institute (MEI), Kansas City, Missouri
  - Washington University, St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Investigators recruited study subjects from their clinic practice. Subjects were randomized to either Group A or Group B at the time of the baseline visit. First patient first visit occurred on May 25, 2012 and last patient last visit occurred on September 07, 2012.
Groups:
- Control First, Then Experimental (Group A): Initial subject use of Control Sound Processing Strategy for the first week, followed by subject use of Experimental Sound Processing Strategy for the HiResolution™ Bionic Ear System for the second week.
  Control Sound Processing Strategy: HiRes Fidelity120™ Sound Processing Strategy, which is currently marketed sound processing strategy.
  Experimental Sound Processing Strategy: newly modified sound processing strategy for the HiResolution™ Bionic Ear System.
- Experimental First, Then Control (Group B): Initial subject use of Experimental Sound Processing Strategy for the first week for the HiResolution™ Bionic Ear System, followed by subject use of Control Sound Processing Strategy for the second week.
  Control Sound Processing Strategy: HiRes Fidelity120™ Sound Processing Strategy, which is currently marketed sound processing strategy.
  Experimental Sound Processing Strategy: newly modified sound processing strategy for the HiResolution™ Bionic Ear System.
Period: Overall Study
Arm/Group | Control First, Then Experimental (Group A) | Experimental First, Then Control (Group B)
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control First, Then Experimental (Group A) | Experimental First, Then Control (Group B) | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (14.81) | 58.9 (13.86) | 60.4 (14.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Speech Perception With Control and Experimental Conditions Both Tested in Quiet, in Speech-spectrum Noise, and in Multi-talker Babble Noise.
Description: Sentence recognition with the new (experimental) and current (control) sound processing strategies will be compared. Subjects will be tested using the AzBio corpus of sentences, which consists of 33 lists of 20 sentences each (6 to 10 words per sentence) that are equated for intelligibility. The difference between the Control percent correct scores and Experimental percent correct scores will be used for the analysis (Experimental AzBio scores minus Control AzBio scores). Data from both Group A and Group B were pooled for the analysis.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Percent Correct
Groups:
- Group A and Group B Data Pooled: Data from Group A (n=18) and Group B (n=18) were pooled for the statistical analyses. Control data consists of Week 1 data from Group A and Week 2 data from Group B; Experimental data consisted of Week 2 data from Group A and Week 1 data from Group B. The resulting mean Control score was subtracted from the mean Experimental score to yield a paired difference score (i.e. Experimental - Control = paired difference score). The paired difference score (n=36) is reported below for each listening condition.
- Control: Data from Group A and Group B were pooled for the statistical analyses. Control data consists of Week 1 data from Group A and Week 2 data from Group B.
- Experimental: Data from Group A and Group B were pooled for the statistical analyses. Experimental data consisted of Week 2 data from Group A and Week 1 data from Group B.
Arm/Group | Group A and Group B Data Pooled | Control | Experimental
Number analyzed (Participants) | 36 | 36 | 36
Percent Correct
  Quiet | 0.2 (6.06) | 88.3 (11.15) | 88.5 (12.43)
  SSN | 2.8 (8.28) | 61.2 (18.98) | 64.0 (18.11)
  MTB | 2.2 (6.89) | 67.8 (17.13) | 70.0 (16.53)

2. Primary Outcome: Device-related Adverse Events
Description: Device-related adverse events will be assessed to determine whether they impact current device safety performance.
Time Frame: 2 weeks
Measure: Number; unit: Events
Arm/Group | Control First, Then Experimental (Group A) | Experimental First, Then Control (Group B)
Number analyzed (Participants) | 18 | 18
Events | 0 | 0

ADVERSE EVENTS:
Groups:
- Control First, Then Experimental (Group A): Initial subject use of Control Sound Processing Strategy for the first week, followed by subject use of Experimental Sound Processing Strategy for the HiResolution™ Bionic Ear System condition for the second week.
  Control Sound Processing Strategy: HiRes Fidelity 120™ Sound Processing Strategy, which is currently marketed sound processing strategy.
  Experimental Sound Processing Strategy: newly modified sound processing strategy for the HiResolution™ Bionic Ear System.
- Experimental First, Then Control (Group B): Initial subject use of Experimental Sound Processing Strategy for the first week for the HiResolution™ Bionic Ear System, followed by subject use of the Control Sound Processing Strategy for the second week.
  Control Sound Processing Strategy: HiRes Fidelity 120™ Sound Processing Strategy, which is currently marketed sound processing strategy.
  Experimental Sound Processing Strategy: newly modified sound processing strategy for the HiResolution™ Bionic Ear System.
Arm/Group | Control First, Then Experimental (Group A) | Experimental First, Then Control (Group B)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 2/18 | 3/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control First, Then Experimental (Group A) (N=18) | Experimental First, Then Control (Group B) (N=18)
Headache (General disorders) | 1 (1) | 3 (3)
Cold (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees to submit any publication to Sponsor (S) at least 30 days prior to submission. Within 30 days of its receipt, S advises PI in writing of any information contained therein which is Confidential Information (CI) (other than Study Data) or which may impair the availability of patent protection for Inventions. S has the right to require PI to remove specifically identified CI and/or to delay the publication for an additional 60 days to enable S to seek patent protection for Inventions.